CLINICAL TRIAL: NCT00890435
Title: A Pharmacokinetic Participation Questionnaire Study
Brief Title: Decision Making About Participating in Pharmacokinetic Studies in Patients Enrolled in a Phase I Treatment Clinical Trial
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ADVL08N1; COG-ADVL08N1 (Other: Children's Oncology Group); NCI-08-C-0223; CDR0000616064 (Other: Clinical Trials.gov)
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2014-02

CONDITIONS: Brain and Central Nervous System Tumors; Leukemia; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific; recurrent childhood brain stem glioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood ependymoma; recurrent childhood pineoblastoma; recurrent childhood subependymal giant cell astrocytoma; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; childhood choroid plexus tumor; childhood craniopharyngioma; childhood ependymoblastoma; childhood medulloepithelioma; childhood meningioma; childhood mixed glioma; childhood oligodendroglioma; adult astrocytic tumors; adult brain stem glioma; adult choroid plexus tumor; adult craniopharyngioma; adult ependymoblastoma; adult medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult ependymal tumors; adult meningeal tumor; adult mixed glioma; adult oligodendroglial tumors; adult pineal parenchymal tumor; recurrent adult brain tumor; relapsing chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary acute myeloid leukemia; acute undifferentiated leukemia; mast cell leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; T-cell large granular lymphocyte leukemia; refractory chronic lymphocytic leukemia; childhood chronic myelogenous leukemia; chronic myelomonocytic leukemia; juvenile myelomonocytic leukemia; refractory hairy cell leukemia; prolymphocytic leukemia
MeSH Terms: conditions — Central Nervous System Neoplasms; Leukemia; Astrocytoma; Medulloblastoma; Familial ependymoma; Optic Nerve Glioma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Choroid Plexus Neoplasms; Meningioma; Oligodendroglioma; Craniopharyngioma; Neuroectodermal Tumors, Primitive; Meningeal Neoplasms; Glioma; Pinealoma; Brain Neoplasms; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Biphenotypic, Acute; Leukemia, Mast-Cell; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Large Granular Lymphocytic; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Myelomonocytic, Juvenile; Leukemia, Hairy Cell; Leukemia, Prolymphocytic | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire administration
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Gathering information about why patients or their guardians agree or decline to participate in the optional pharmacokinetic portion of a phase I treatment study may help doctors plan clinical trials in the future.

PURPOSE: This clinical trial is looking at decision making about participating in pharmacokinetic studies in patients enrolled in a phase I treatment clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* To use a simple 2-page survey to gather preliminary information on why patients or parents/guardians (if patient is a minor) do or do not agree to participate in the optional pharmacokinetic portion of a phase I treatment study while consenting to participate in the phase I treatment study.

OUTLINE: This is a multicenter study.

Patients or parents/guardians (if patient is a minor) complete a short questionnaire on the reasons for agreeing/declining to participation in the optional pharmacokinetic sampling component of the phase I clinical trial.

Patient demographics and other relevant information are collected.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients or their parents/guardians (if patient is a minor) consented to participate in a phase I treatment clinical trial with an optional pharmacokinetic (PK) component, within the past 4 weeks

  * Must not have withdrawn consent for the phase I treatment study

    * Patients or their parents/guardians are eligible regardless of whether they initially agreed to participate in the PK sampling

      * Must not withdraw consent for PK sampling prior to completing the study questionnaire if initially agreed to optional PK sampling
    * Patients or their parents/guardians are eligible regardless of whether they actually completed PK sampling (provided reasons for not completing the sampling was not withdrawal of the initial consent to the phase I treatment study)

PATIENT CHARACTERISTICS:

* Not cognitively or physically impaired
* May participate no more than once in the study questionnaire survey

PRIOR CONCURRENT THERAPY:

* No limit on participation in the number of prior phase I trials or other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A patient (family) who has consented to participate in a Phase I trial.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Correlation between study questionnaire answers and patient demographics | Length of study
Correlation between study questionnaire answers and time required by pharmacokinetic sampling | Length of study
Correlation between study questionnaire answers and the need for additional IV | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Fox, MD, Principal Investigator — National Cancer Institute (NCI)